CLINICAL TRIAL: NCT03258593
Title: A Phase I Single-Arm Study of the Combination of Durvalumab (MEDI4736) and Vicineum (Oportuzumab Monatox, VB4-845) in Subjects With High-Grade Non-Muscle-Invasive Bladder Cancer Previously Treated With Bacillus Calmette-Guerin (BCG)
Brief Title: Durvalumab and Vicineum in Subjects With High-Grade Non-Muscle-Invasive Bladder Cancer Previously Treated With Bacillus Calmette-Guerin (BCG)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Raju Chelluri, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 170157; 17-C-0157
Record Dates: First submitted 2017-08-22; First posted 2017-08-23 (Actual); Results first posted 2023-10-26 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Urinary Bladder Neoplasms
Keywords: Carcinoma-in-situ; High-grade Ta or T1 disease; Papillary Tumors
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma in Situ | interventions — durvalumab; Acetaminophen; Histamine Antagonists; Diphenhydramine; Cystoscopy; Electrocardiography; Tomography, X-Ray Computed; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg (Experimental): Durvalumab + Vicineum, escalating doses. Up to 2 dose levels will be evaluated in the first 6 - 12 participants.
  Interventions: Drug: Durvalumab; Drug: Vicineum; Drug: Acetaminophen; Drug: Antihistamine; Procedure: Bladder Biopsy; Procedure: TURBT; Procedure: Cystoscopy; Diagnostic Test: Urine cytology; Diagnostic Test: Electrocardiogram; Diagnostic Test: CT; Diagnostic Test: MRI
- Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg (Experimental): Durvalumab + Vicineum, at the maximum tolerated dose (MTD). Up to 24 participants.
  Interventions: Drug: Durvalumab; Drug: Vicineum; Drug: Acetaminophen; Drug: Antihistamine; Procedure: Bladder Biopsy; Procedure: TURBT; Procedure: Cystoscopy; Diagnostic Test: Urine cytology; Diagnostic Test: Electrocardiogram; Diagnostic Test: CT; Diagnostic Test: MRI
- Level 1, Durvalumab 1500mg intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 20 mg (Experimental): Level 1, Durvalumab 1500mg intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 20 mg
  Interventions: Drug: Durvalumab; Drug: Vicineum; Drug: Acetaminophen; Drug: Antihistamine; Procedure: Bladder Biopsy; Procedure: TURBT; Procedure: Cystoscopy; Diagnostic Test: Urine cytology; Diagnostic Test: Electrocardiogram; Diagnostic Test: CT; Diagnostic Test: MRI
- Arm 2, Durvalumab + Vicineum at the Maximum Tolerated Dose (MTD) (Experimental): Arm 2, Durvalumab + Vicineum at the Maximum Tolerated Dose (MTD)
  Interventions: Drug: Durvalumab; Drug: Vicineum; Drug: Acetaminophen; Drug: Antihistamine; Procedure: Bladder Biopsy; Procedure: TURBT; Procedure: Cystoscopy; Diagnostic Test: Urine cytology; Diagnostic Test: Electrocardiogram; Diagnostic Test: CT; Diagnostic Test: MRI

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 1500 mg is administered intravenously (IV) once every 4 weeks for 12 months with an option to continue therapy for an additional 12 months (total of 24 months) provided that, participant is tolerating therapy and remains free of recurrent high grade NMIBC (see Treatment Period below). The dose of durvalumab is 1500 mg. If optional maintenance therapy continued in the second year, durvalumab 1500 mg will be administered intravenously once every 3 months to provide an immune boost.
  Other Names: Imfinzi
Drug: Vicineum — Vicineum is administered in a 12-week Induction Phase followed by a Maintenance Phase for at least one year with an option for a total of up to 2 years of treatment. During the Induction Phase, Vicineum is administered once weekly for 12 weeks. During the Maintenance Phase, Vicineum is administered every other week. The dose of Vicineum is 30 mg in 50 mL of saline.
Drug: Acetaminophen — Acetaminophen or equivalent medications per institutional standard may be administered at the discretion of the investigator.
  Other Names: Tylenol; Panadol; Paracetamol
Drug: Antihistamine — Antihistamine (e.g., diphenhydramine) or equivalent medications per institutional standard may be administered at the discretion of the investigator.
  Other Names: Diphenhydramine
Procedure: Bladder Biopsy — Bladder biopsy at screening and every 3 months before each cystoscopy per schema.
Procedure: TURBT — Transurethral resection of a bladder tumor (TURBT) at screening and every 3 months before each cystoscopy per schema.
  Other Names: Transurethral resection of a bladder tumor
Procedure: Cystoscopy — Urine cytology at screening and every 3 months before each cystoscopy per schema.
Diagnostic Test: Urine cytology — Urine cytology at baseline and every 3 months before each cystoscopy per schema.
Diagnostic Test: Electrocardiogram — Electrocardiogram (ECG) at screening, pre-durvalumb infusion and as clinically indicated during the trial.
  Other Names: ECG
Diagnostic Test: CT — Computed tomography (CT) at screening and every 12 months while on study.
  Other Names: Computed tomography
Diagnostic Test: MRI — Magnetic resonance imaging (MRI) at screening and every 12 months while on study.
  Other Names: Magnetic resonance imaging

SUMMARY:
Background:

Non-muscle-invasive bladder cancer is in the early stages. But it usually comes back after treatment. The drugs Vicineum and Durvalumab may help the immune system find and destroy cancer cells.

Objective:

To test if the drugs Durvalumab and Vicineum together are safe and effective to treat people with bladder cancer that has not spread to the muscle in the bladder.

Eligibility:

People ages 18 and older who have bladder cancer that has not spread to the muscle in the bladder and was treated unsuccessfully with Bacillus Calmette-Guerin

Design:

Participants will be screened with:

Medical history

Physical exam

Blood and urine tests

Tumor sample from previous surgery. If one is not available, they will have a biopsy: A small piece of tumor is removed.

Cystoscopy to examine the inside of the bladder. This may include a biopsy or removing tumors.

Computed tomography (CT) or magnetic resonance imaging (MRI): They lie in a machine that takes pictures of the body.

Electrocardiogram to test heart function

Participants will receive Durvalumab and Vicineum in 2 phases:

First phase: Durvalumab every 4 weeks and Vicineum once a week for 3 months

Second phase: Durvalumab every 4 weeks and Vicineum once every other week

Participants will have tumor samples taken every 3 months. They will have blood and urine tests throughout the study.

Participants will continue treatment for up to 2 years.

Participants will have a visit about 30 days after their last treatment. This includes blood and urine tests. It may include a cytoscopy or additional biopsies.

DETAILED DESCRIPTION:
In 2016, it is estimated that there will be 76,960 new cases of bladder cancer and 16,390 deaths associated with bladder cancer. Bladder cancer is associated with the highest costs among all types of cancer, due to the need for lifelong routine monitoring and treatment. Approximately 70% of cases are non-muscle invasive bladder cancer (NMIBC) at presentation and are treated by transurethral resection of bladder tumor (TURBT) followed by intravesical treatment with BCG (Bacillus Calmette-Guerin) or mitomycin C. However, in the setting of high-grade disease, these therapies can become ineffective over time in up to two-thirds of patients and disease progression to muscle invasive bladder cancer (MIBC) can occur. In patients who present with CIS (carcinoma in situ) rates of progression are greater than 50%. Progression to MIBC portends a poor outcome as only 50% of patients will survive five years despite undergoing radical cystectomy. Clearly, there is a large unmet need in therapeutic options for NMIBC that recurs or progresses.

Vicineum(TM) is a recombinant fusion protein, VB4-845, that contains a humanized single-chain antibody fragment specific for the epithelial cell adhesion molecule (EpCAM) antigen linked to ETA (252-608), a truncated form of Pseudomonas exotoxin A (ETA). EpCAM is overexpressed on the surface of urothelial carcinoma cells and therefore represents a good target for Vicineum(TM) to bind to. In a previous phase II study in BCG refractory or BCG intolerant patients with high grade bladder cancer, 16% of patients treated with induction and maintenance therapy with Vicineum(TM) remained disease-free at 1 year. As a result, Vicineum(TM) is currently being evaluated as a single agent in a phase III trial.

Pre-clinical work with a drug called Proxinium, an earlier version of Vicineum(TM), demonstrated an abscopal effect and synergy with the use of a checkpoint blockade inhibitor. Although it was done in a non-small cell lung cancer (NSCLC) model, the results were impressive in causing tumor shrinkage. Durvalumab is a human monoclonal antibody (MAb) that inhibits binding of programmed cell death ligand 1 (PD-L1) (B7 homolog 1 [B7-H1], cluster of differentiation [CD]274) to programmed cell death 1 (PD-1; CD279) and CD80 (B7-1). Durvalumab has been demonstrated to have activity against advanced metastatic urothelial bladder cancer whose tumor has progressed during or after one standard platinum-based regimen in a phase I trial.

Therefore, this trial will take two agents with single agent activity against urothelial cancer and combine them in a Phase I trial for patients with high-grade NMIBC Previously Treated with BCG.

Objectives:

Primary Objectives:

To evaluate the safety and tolerability of durvalumab and Vicineum when administered in combination to subjects with BCG-refractory high-grade NMIBC

Eligibility:

Subjects must have a histologically confirmed high-grade non-muscle invasive urothelial carcinoma (transitional cell carcinoma) of the bladder as follows:

Carcinoma-in-situ (CIS) with or without papillary tumors

High-grade Ta or T1 disease based on a biopsy/TURBT performed within 12 weeks of the initial dose of study treatment. If multiple bladder biopsies/TURBTs are required to confirm eligibility, the timing of the last bladder biopsy to the initial dose of study treatment must be within 12 weeks.

Subjects with BCG unresponsive disease as defined by the Society of Urologic Oncology and the Food and Drug Administration (FDA): Subjects must have received at least two courses of intravesical BCG (at least 5 of 6 induction doses of BCG and at least 2 of 3 maintenance doses of BCG under a maintenance regimen or at least 2 doses of a repeat induction course). See exception below for persistent T1 disease below. There is no upper limit on the amount of prior BCG a subject may have received.

Patients with persistent T1 high grade disease on TURBT following a single induction course of BCG (at least 5 of 6 doses) may also be eligible for this trial provided that the patient is surgically unfit for cystectomy as deemed by the investigator or the patient declines cystectomy

Design:

This is a Phase I, open-label study of the combination of durvalumab and Vicineum in subjects with high-grade NMIBC previously treated with BCG.

All subjects will receive Vicineum intravesically and durvalumab systemically at the standard doses for both drugs as determined by Phase II trials for each drug, as no synergy or additive effect is expected for adverse events.

Vicineum is administered in a 12-week Induction Phase followed by a Maintenance Phase for at least one year with an option for a total of up to 2 years of treatment. During the Induction Phase, Vicineum is administered once weekly for 12 weeks. During the Maintenance Phase, Vicineum is administered every other week. The dose of Vicineum is 30 mg in 50 mL of saline.

Durvalumab 1500 mg is administered intravenously (IV) once every 4 weeks for 12 months with an option to continue therapy for an additional 12 months (total of 24 months) provided that patient is tolerating therapy and remains free of recurrent high grade NMIBC (see Treatment Period below). The dose of durvalumab is 1500 mg. If optional maintenance therapy continued in the second year, durvalumab 1500 mg will be administered intravenously once every 3 months to provide an immune boost.

Vicineum will be given as monotherapy for 1 week followed by treatment with the combination of Vicineum and durvalumab starting week 2.

In the initial six patients, three subjects at a time will enroll at these doses and schedules. Dose-liming toxicity (DLT) for each subject will be determined during the initial 6-week period that the subject is on treatment (i.e., the DLT period). When all subjects in the initial cohort have been on treatment through the DLT period, all available safety data will be considered in decisions to enroll additional subjects at this dose level, or to de-escalate the dose(s) of study drug(s), based on a standard "3 + 3" design. There will be no dose-escalations in this study. The dose of durvalumab will remain at 1500 mg every 4 weeks, and the dose of each intravesical Vicineum treatment can be reduced to 20 mg if the initial doses in combination induce DLTs.

After the first six patients, an additional 18 subjects will be enrolled at the initial doses or at the reduced doses (if DLTs resulted in the first 6 patients) in order to obtain additional safety data, biomarker data and preliminary anti-tumor activity.

Each subject's course will consist of the following periods:

Screening/Baseline Period: The subject is consented and undergoes screening assessments to determine eligibility for the study.

Treatment Period: The subject is treated and monitored for safety. Biomarker data will be obtained prior to treatment and at periodic intervals during treatment. Subjects who remain free of high-grade NMIBC after 12 months of study treatment may continue to receive treatment for an additional 12 months until they develop recurrent high-grade disease, disease progression, or intolerable toxicity, or meet another withdrawal criterion (e.g., consent withdrawal, pregnancy).

Post-Treatment. The subject will return to the study site monthly for up to 90 days after the last dose of immunotherapy for end-of-treatment assessments. Subjects with ongoing clinically significant related adverse events (AEs) or serious adverse events (SAEs) will have additional follow-up after the initial post-treatment visit.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically or cytologically confirmed by National Cancer Institute (NCI) Laboratory of Pathology as high-grade non-muscle invasive urothelial (transitional cell carcinoma) of the bladder as follows:

  * Carcinoma-in-situ (CIS) with or without papillary tumors
  * High-grade Ta or T1 disease based on a biopsy/transurethral resection of bladder tumor (TURBT) performed within 12 weeks of the initial dose of study treatment. If multiple bladder biopsies/TURBTs are required to confirm eligibility, the timing of the last bladder biopsy to the initial dose of study treatment must be within 12 weeks.
  * Patients with persistent T1 high grade disease on TURBT following a single induction course of BCG (Bacillus Calmette-Guerin) (at least 5 of 6 doses) may also be eligible for this trial provided that the patient is surgically unfit for cystectomy as deemed by the investigator or the patient declines cystectomy.
* Subjects with BCG unresponsive disease as defined by the Society of Urologic Oncology and the Food and Drug Administration (FDA): Subjects must have received at least two courses of intravesical BCG (at least 5 of 6 induction doses of BCG and at least 2 of 3 maintenance doses of BCG under a maintenance regimen or at least 2 doses of a repeat induction course). Please note exception above for persistent T1 disease. There is no upper limit on the amount of prior BCG a subject may have received.
* Patients who have met eligibility criterion above must have received last BCG dose within a year of enrollment.
* The investigator must document that he/she believes the subject would not benefit from additional BCG treatment at the time of study entry.
* Age >= 18 years at time of signing the informed consent form (ICF). Because no dosing or adverse event data are currently available on the use of Vicineum in combination with durvalumab in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials. Furthermore, non-muscle invasive bladder cancer (NMIBC) does not occur in children.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate organ and marrow function as defined below:

  * Hemoglobin >= 9.0 g/dL
  * Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (> 1500 per mm^3)
  * Platelet count >= 75 x 10^9/L (>75,000 per mm^3)
  * Serum bilirubin less than or equal to 1.5 x institutional upper limit of normal (ULN).
  * Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamate-pyruvate transaminase (SGPT) less than or equal to 2.5 x institutional ULN
  * Creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

    * Males: Creatinine CL (mL/min) = (Weight (kg) x (140 - Age))/72 x serum creatinine (mg/dL)
    * Females: Creatinine CL (mL/min) = (Weight (kg) x (140 - Age) x 0.85)/72 x serum creatinine (mg/dL)
* Female subjects must either be of non-reproductive potential (i.e., post-menopausal as described below) OR history of surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.

  * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution
  * Women >= 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, or had chemotherapy-induced menopause with last menses >1 year ago
* The effects of Vicineum and durvalumab on the developing human fetus are unknown. For this reason, all sexually active subjects agree to use barrier contraception (i.e., condoms) while receiving study treatment and for 120 days following their last dose of study treatment. Female subjects of child-bearing potential and male subjects whose sexual partners are women of childbearing potential (WOCBP) agree to use barrier contraception and a second form of contraception while receiving study treatment and for 4 months following their last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Written informed consent obtained from the subject prior to performing any protocol- related procedures
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Body weight > 30 kg

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents.
* QT interval corrected for heart rate using Fridericia's formula the corrected QT interval by Fridericia (QTcF) >=470 ms. (Any clinically significant abnormalities detected require triplicate ECG results and a mean QT interval corrected for heart rate using Fridericia's formula (QTcF) >=470 ms calculated from 3 ECGs.)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Vicineum or durvalumab or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Urinary tract infections (UTIs) are excluded from being an exclusion criterion for treatment unless they are grade 3 or higher.
* Pregnant women are excluded from this study because it is unknown whether Vicineum and/or durvalumab have any teratogenic effects. In nursing mothers, breastfeeding should be discontinued as these medications may have the potential risk for adverse events in nursing infants secondary to treatment of the mother.
* Any previous treatment with a programmed cell death 1 (PD-1) or programmed death-ligand 1 (PD-L1) inhibitor, including durvalumab
* Evidence of non-bladder urothelial (transitional cell) carcinoma by biopsy, cytology, or radiological imaging within the past 2 years of treatment (e.g., upper tract transitional cell carcinoma, urethral urothelial carcinoma).
* Subjects with hydronephrosis, except for those subjects where hydronephrosis has been longstanding (i.e., predates the diagnosis of the CIS (carcinoma in situ), Ta, or T1 by more than 2 years) and diagnostic evaluation at screening shows no evidence of tumor causing the hydronephrosis.
* Any other anticancer therapy (e.g., chemotherapy, biologic therapy, immunotherapy, targeted therapy, endocrine therapy, radiation therapy, intravesical therapy, investigational agent) within 28 days of the first dose of study therapy (and within 6 weeks for nitrosourea or mitomycin C) other than a single dose of intravesical chemotherapy which is permitted between 28 days and 14 days prior to the first dose of study treatment.
* The subject has a diagnosis of another malignancy within 2 years before the first dose of study treatment, except for superficial skin cancer, localized prostate cancer on active surveillance, or localized solid tumors deemed cured by surgery and not treated with systemic anticancer therapy and not expected to require anticancer therapy in the next 2 years i.e., while the subject may be taking study treatment.
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Grave's disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

  * Subjects with vitiligo or alopecia
  * Subjects with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormonal replacement
  * Any chronic skin condition that does not require systemic therapy
  * Subjects without active disease in the last 5 years may be included but only after consultation with the Principal Investigator
  * Subjects with celiac disease controlled by diet alone
* History of primary immunodeficiency.
* History of allogeneic organ transplant.
* History of hypersensitivity to durvalumab or any excipient
* History of hypersensitivity to Vicineum or its components
* Active infection with tuberculosis (clinical evaluation that includes clinical history, physical examination, and radiographic findings, and purified protein derivative (PPD) testing if indicated), hepatitis B (known positive HBV surface antigen (HBsAg) result, hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with HIV are excluded from participating on this clinical trial because their immunodeficiency would confound the evaluation of adverse events which would hinder meeting the primary objective. Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA).
* History of leptomeningeal carcinomatosis
* Receipt of live attenuated vaccination within 30 days prior to the first dose of Vicineum or durvalumab
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
* Subjects with uncontrolled seizures
* Any unresolved toxicity National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade >=2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

  * Subjects with Grade >=2 neuropathy will be evaluated on a case-by-case basis after consultation with the Principal Investigator.
  * Subjects with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Principal Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raju Chelluri, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol genomic data sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0157.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled in Level 1, Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 20 mg, and Arm 2, Durvalumab + Vicineum at the Maximum Tolerated Dose (MTD).
Groups:
- Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg: Durvalumab 1500 mg is administered intravenously (IV) once every 4 weeks for 12 months with an option to continue therapy for an additional 12 months (total of 24 months) provided that, participant is tolerating therapy and remains free of recurrent high grade non-muscle invasive bladder cancer (NMIBC) (see Treatment Period below). The dose of durvalumab is 1500 mg. If optional maintenance therapy continued in the second year, durvalumab 1500 mg will be administered intravenously once every 3 months to provide an immune boost.
  Vicineum is administered in a 12-week Induction Phase followed by a Maintenance Phase for at least one year with an option for a total of up to 2 years of treatment. During the Induction Phase, Vicineum is administered once weekly for 12 weeks. During the Maintenance Phase, Vicineum is administered every other week. The dose of Vicineum is 30 mg in 50 mL of saline.
- Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg: Durvalumab + Vicineum, at the maximum tolerated dose (MTD). Durvalumab: an option to continue therapy for an additional 12 months (total of 24 months) provided that, participant is tolerating therapy and remains free of recurrent high grade NMIBC (see Treatment Period below). The dose of durvalumab is 1500 mg. If optional maintenance therapy continued in the second year, durvalumab 1500 mg will be administered intravenously once every 3 months to provide an immune boost.
  Vicineum is administered in a 12-week Induction Phase followed by a Maintenance Phase for at least one year with an option for a total of up to 2 years of treatment. During the Induction Phase, Vicineum is administered once weekly for 12 weeks. During the Maintenance Phase, Vicineum is administered every other week. The dose of Vicineum is 30 mg in 50 mL of saline.
- Level 1, Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 20 mg: Durvalumab 1500 mg is administered intravenously (IV) once every 4 weeks for 12 months with an option to continue therapy for an additional 12 months (total of 24 months) provided that, participant is tolerating therapy and remains free of recurrent high grade NMIBC (see Treatment Period below). The dose of durvalumab is 1500 mg. If optional maintenance therapy continued in the second year, durvalumab 1500 mg will be administered intravenously once every 3 months to provide an immune boost.
  Vicineum is administered in a 12-week Induction Phase followed by a Maintenance Phase for at least one year with an option for a total of up to 2 years of treatment. During the Induction Phase, Vicineum is administered once weekly for 12 weeks. During the Maintenance Phase, Vicineum is administered every other week. The dose of Vicineum is 20mg in 50 mL of saline
- Arm 2, Durvalumab + Vicineum at the Maximum Tolerated Dose (MTD): Durvalumab 1500 mg is administered intravenously (IV) once every 4 weeks for 12 months with an option to continue therapy for an additional 12 months (total of 24 months) provided that, participant is tolerating therapy and remains free of recurrent high grade NMIBC (see Treatment Period below). The dose of durvalumab is 1500 mg. If optional maintenance therapy continued in the second year, durvalumab 1500 mg will be administered intravenously once every 3 months to provide an immune boost.
  Vicineum is administered in a 12-week Induction Phase followed by a Maintenance Phase for at least one year with an option for a total of up to 2 years of treatment. During the Induction Phase, Vicineum is administered once weekly for 12 weeks. During the Maintenance Phase, Vicineum is administered every other week. The dose of Vicineum is 30 mg in 50 mL of saline
Period: Run-In Induction Phase
Arm/Group | Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Level 1, Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 20 mg | Arm 2, Durvalumab + Vicineum at the Maximum Tolerated Dose (MTD)
Started | 12 | 0 | 0 | 0
Completed | 12 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Run-In Maintenance Phase
Arm/Group | Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Level 1, Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 20 mg | Arm 2, Durvalumab + Vicineum at the Maximum Tolerated Dose (MTD)
Started | 12 | 0 | 0 | 0
Completed | 5 | 0 | 0 | 0
Not Completed | 7 | 0 | 0 | 0
Not completed — Disease recurrence | 4 | 0 | 0 | 0
Not completed — Disease progression | 3 | 0 | 0 | 0
Period: Expansion Induction Phase
Arm/Group | Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Level 1, Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 20 mg | Arm 2, Durvalumab + Vicineum at the Maximum Tolerated Dose (MTD)
Started | 0 | 3 | 0 | 0
Completed | 0 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Expansion Maintenance Phase
Arm/Group | Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Level 1, Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 20 mg | Arm 2, Durvalumab + Vicineum at the Maximum Tolerated Dose (MTD)
Started | 0 | 3 | 0 | 0
Completed | 0 | 1 | 0 | 0
Not Completed | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Total
Number analyzed (Participants) | 12 | 3 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 10 | 2 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (8) | 72 (10) | 72 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 11 | 3 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 3 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 2 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Grades 1-5 Adverse Events
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. Grade 1 is mild, grade 2 is moderate, grade 3 is severe, grade 4 is life-threatening, and grade 5 is death related to adverse event.
Time Frame: Through study completion, an average of 315 days
Measure: Number; unit: adverse events
Groups:
- Total Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg: Total Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg
Arm/Group | Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Total Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg
Number analyzed (Participants) | 12 | 3 | 15
adverse events
  Grade 1 | 12 | 3 | 15
  Grade 2 | 9 | 3 | 12
  Grade 3 | 4 | 0 | 4
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

2. Secondary Outcome: Urinary Epithelial Cell Adhesion Molecule (EpCAM) Compared Between Participants Who Have a Clinical Response to Therapy vs. Those Who do Not Respond
Description: Urinary EpCAM will be measured and will be compared between participants who have a clinical response to therapy vs. those who do not respond. Although it is expected to have low power, a comparison of the EpCAM levels may be compared between the two response categories using a Wilcoxon rank sum test, with the resulting p-value intended to help describe the differences noted.
Time Frame: Baseline, week 1, weeks 2-5, week 6, week 10 and week 12
Reporting Status: Not Posted, anticipated posting 2026-02

3. Secondary Outcome: Response Rate
Description: The response to treatment will be determined for evaluable participants who receive treatment and was measured as follows: Recurrence is suspected and/or determined by urine cytology and/or cystoscopic exam and then confirmed pathologically after a transurethral resection of bladder tumor (TURBT). Complete response rate for carcinoma in situ (CIS) is defined as the absence of CIS upon follow-up biopsies. Disease progression is defined as upstaging from a lower stage to a higher stage (e.g., Ta to T1-T4 or T1 to T2-4; CIS to T1 or CIS to T2-T4; or any N+ or M+ in these high-grade tumors).
Time Frame: From enrollment until event occurrence (recurrence, progression); twelve weeks.
Measure: Number; unit: percentage of participants
Arm/Group | Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Total Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg
Number analyzed (Participants) | 12 | 3 | 15
percentage of participants
  Complete response | 41.6 | 66.6 | 46.6
  Recurrence | 58.3 | 33.3 | 53.3
  Disease progression | 25 | 33.3 | 26.6

4. Secondary Outcome: Pharmacokinetic Parameters in Urine Maximum Concentration (Cmax) of Vicineum
Description: Evaluate the pharmacokinetic parameters of Vicineum obtained by urine samples. Urinary Vicineum (in ng/mL).
Time Frame: Baseline, week 1, week 6, week 12
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Total Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg
Number analyzed (Participants) | 12 | 3 | 15
ng/mL
  Baseline | 2.5 [1.5 to 3.8] | 1.5 [1.5 to 1.5] | 3.2 [2.1 to 7.4]
  Week 1, Day 1 | 4320.0 [10.6 to 11965.5] | 305.4 [195.8 to 15231.8] | 3738.7 [49.9 to 14072.6]
  Week 1 | 2.6 [1.7 to 5.5] | 1.5 [1.5 to 1.5] | 4.7 [2.1 to 6.5]
  Week 6 | 3.2 [1.5 to 4.7] | 1.5 [1.5 to 1.5] | 4.3 [2.4 to 7.5]
  Week 12 | 3.5 [1.8 to 5.5] | 7.5 [7.5 to 7.5] | 4.8 [2.1 to 7.5]

5. Secondary Outcome: Change in Programmed Death-ligand 1 (PD-L1) Levels Between Responders and Non-Responders
Description: PD-L1 levels will be obtained at baseline and after treatment with both agents. The change in levels will be determined between the two measurements, and these changes will be compared between responders and non-responders. Although it is expected to have low power, in each case the comparisons between the two response categories will be made using a Wilcoxon rank sum test, with the resulting p-value intended to help describe the differences noted.
Time Frame: Baseline and after treatment with both agents, from enrollment up to 5 weeks
Population: Number of responders and non-responders in the rows below = overall number of participants analyzed for each group.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Total Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg
Number analyzed (Participants) | 12 | 3 | 15
pg/mL
  Responders PDL1 levels after treatment (vs baseline: number analyzed (Participants) | 5 | 2 | 7
  Responders PDL1 levels after treatment (vs baseline | 573.4 [533.8 to 670.3] | 342.5 [319.4 to 365.6] | 533.8 [443.5 to 621.8]
  Non-responders PDL1 levels after treatment (vs baseline): number analyzed (Participants) | 7 | 1 | 8
  Non-responders PDL1 levels after treatment (vs baseline) | 505.9 [421.3 to 532.4] | 228.4 [228.4 to 228.4] | 489.7 [368.6 to 524.2]
Statistical Analysis 1: Comparison: Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg; Test type: Other — Location Tests (Wilcoxon Rank sum test); p = 0.202, Wilcoxon Rank sum test — Unadjusted p-value; Median Difference (Net) = 67.5, 95% CI 2-sided [25 to 75]
Statistical Analysis 2: Comparison: Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg; Test type: Other — Location Tests (Wilcoxon Rank sum test); p = 0.667, Wilcoxon Rank sum test — Unadjusted p-value; Median Difference (Net) = 114, 95% CI 2-sided [67.9 to 160.3]
Statistical Analysis 3: Comparison: Total Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg; Test type: Other — Location Tests (Wilcoxon Rank sum test); p = 0.463, Wilcoxon Rank sum test; Median Difference (Net) = 44.1, 95% CI 2-sided [25 to 75]

6. Secondary Outcome: Change in Programmed Cell Death Protein 1 (PD-1) Levels Between Responders and Non-Responders
Description: PD-1 levels will be obtained at baseline and after treatment with both agents. The change in levels will be determined between the two measurements, and these changes will be compared between responders and non-responders. Although it is expected to have low power, in each case the comparisons between the two response categories will be made using a Wilcoxon rank sum test, with the resulting p-value intended to help describe the differences noted.
Time Frame: baseline and after treatment with both agents
Reporting Status: Not Posted, anticipated posting 2026-02

7. Secondary Outcome: Change in Programmed Death-ligand 1 (PD-L1) Levels Between Participants Who Respond and Have Stable Disease (SD), and Those With Progressive Disease (PD)
Description: PD-L1 levels will be obtained at baseline and after treatment with both agents. The change will be compared between those who respond or have stable disease (SD (clinical benefit=Complete Response (CR)+Partial Response (PR)+SD) and those with progressive disease (PD). Although it is expected to have low power, in each case the comparisons between the two response categories will be made using a Wilcoxon rank sum test, with the resulting p-value intended to help describe the differences noted.
Time Frame: Baseline and after treatment, from enrollment up to 5 weeks
Population: Number of participants with SD and participants with PD in the rows below = overall number of participants analyzed for each group.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Total Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg
Number analyzed (Participants) | 12 | 3 | 15
pg/mL
  PDL1 level changes in participants with SD (treatment vs baseline): number analyzed (Participants) | 9 | 2 | 11
  PDL1 level changes in participants with SD (treatment vs baseline) | 533.8 [498.3 to 573.4] | 342.5 [319.4 to 365.6] | 505.9 [378.9 to 561.0]
  PDL1 level changes in participants with PD (treatment vs baseline: number analyzed (Participants) | 3 | 1 | 4
  PDL1 level changes in participants with PD (treatment vs baseline | 516 [494.8 to 612.9] | 228.4 [228.4 to 228.4] | 494.8 [412.2 to 564.6]
Statistical Analysis 1: Comparison: Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg; Test type: Other — Location test (Rank sum based i.e., Wilcoxon test); p = 0.863, Wilcoxon Rank sum test; Median Difference (Net) = -17.75, 95% CI 2-sided [-211.6 to 170.3] — Median change; Signed Rank (S/R) of post-treatment PDL-1 levels minus baseline
Statistical Analysis 2: Comparison: Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg; Test type: Other — Location test (Rank sum based i.e., Wilcoxon test); p = 0.666, Wilcoxon Rank sum test; Median Difference (Net) = 114.1, 95% CI 2-sided [67.9 to 160.3] — Median change; Signed Rank (S/R) of post-treatment PDL-1 levels minus baseline
Statistical Analysis 3: Comparison: Total Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg; Test type: Other — Location test (Rank sum based i.e., Wilcoxon test); p = 0.949, Wilcoxon Rank sum test; Median Difference (Net) = 21.3, 95% CI 2-sided [-203.9 to 269.9] — Median change; Signed Rank (S/R) of post-treatment PDL-1 levels minus baseline

8. Secondary Outcome: Change in Programmed Cell Death Protein 1(PD-1) Levels Between Participants Who Respond and Have Stable Disease (SD), and Those With Progressive Disease (PD)
Description: PD-1 levels will be obtained at baseline and after treatment with both agents. The change will be compared between those who respond or have stable disease (SD (clinical benefit=Complete Response (CR)+Partial Response (PR)+SD) and those with progressive disease (PD). Although it is expected to have low power, in each case the comparisons between the two response categories will be made using a Wilcoxon rank sum test, with the resulting p-value intended to help describe the differences noted.
Time Frame: baseline and after treatment
Reporting Status: Not Posted, anticipated posting 2026-02

9. Secondary Outcome: Changes in the Immune Parameters Obtained From Blood Samples
Description: All evaluable participants will have determinations of many immune parameters at baseline, 3 months, and 6 months. The changes in the parameters obtained from blood samples will be determined at baseline vs. 3 months, and baseline vs. 6 months. Comparisons of the paired values will be performed using a Wilcoxon signed rank test, and a Hochberg adjustment may be used.
Time Frame: baseline, 3 weeks, and 5 weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Total Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg
Number analyzed (Participants) | 12 | 3 | 15
pg/mL
  3 weeks Interferon Gamma (IFN-γ) vs Baseline | 4.340 [0.950 to 9.315] | 0.640 [-0.035 to 2.225] | 3.850 [0.720 to 6.525]
  5 weeks Interferon Gamma (IFN-γ) vs Baseline | 3.290 [1.375 to 8.312] | 1.750 [0.985 to 12.265] | 3.120 [1.370 to 10.825]
  3 weeks Interleukin 6 (IL-6) vs Baseline | 0.395 [0.037 to 0.802] | 0.180 [0.115 to 0.320] | 0.280 [0.050 to 0.590]
  5 weeks Interleukin 6 (IL-6) vs Baseline | 0.540 [-0.070 to 0.870] | 0.220 [0.145 to 0.520] | 0.400 [0.005 to 0.770]
  3 weeks Interleukin 8 (IL-8) vs Baseline | 0.730 [-0.482 to 1.370] | 0.880 [-0.795 to 10.295] | 0.860 [-0.895 to 1.610]
  5 weeks Interleukin 8 (IL-8) vs Baseline | -0.395 [-0.647 to 0.597] | -0.160 [-0.455 to 10.145] | -0.180 [-0.665 to 0.715]
  3 weeks Interleukin 10 (IL-10) vs Baseline | 0.120 [0.047 to 0.202] | 0.07 [-0.04 to 0.15] | 0.120 [0.045 to 0.205]
  5 weeks Interleukin 10 (IL-10) vs Baseline | 0.105 [0.047 to 0.365] | 0.120 [0.075 to 0.305] | 0.120 [0.045 to 0.380]
  3 weeks Tumor Necrosis Factor Alpha (TNF-α) vs Baseline | 0.400 [0.207 to 0.560] | 0.260 [0.100 to 0.525] | 0.350 [0.165 to 0.590]
  5 weeks Tumor Necrosis Factor Alpha (TNF-α) vs Baseline | 0.240 [0.122 to 1.207] | 0.270 [0.175 to 0.320] | 0.270 [0.110 to 0.930]
Statistical Analysis 1: Comparison: Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg vs Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg; Interferon Gamma (IFN-γ) at 3 weeks compared to their respective baseline values; Test type: Other — Other: median difference; p < 0.001, Paired samples Wilcoxon rank sum test — Hochberg adjustment may be used; Median Difference (Net) = 4.34, 95% CI 2-sided [1.7 to 38.0]
Statistical Analysis 2: Comparison: Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg vs Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg; Interferon Gamma (IFN-γ) at 5 weeks compared to their respective baseline values; Test type: Other — Other: median difference; p < 0.001, Paired samples Wilcoxon rank sum test — Hochberg adjustment may be used; Median Difference (Net) = 3.29, 95% CI 2-sided [1.5 to 11.25]
Statistical Analysis 3: Comparison: Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg vs Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg; Tumor Necrosis Factor Alpha (TNF-α) at 3 weeks compared to their respective baseline values; Test type: Other — Other: median difference; p < 0.05, Paired samples Wilcoxon rank sum test — Hochberg adjustment may be used; Median Difference (Net) = 0.4, 95% CI 2-sided [0.1 to 0.7]
Statistical Analysis 4: Comparison: Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg vs Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg; Tumor Necrosis Factor Alpha (TNF-α ) at 5 weeks compared to their respective baseline values; Test type: Other — Other: median difference; p = 0.052, Paired samples Wilcoxon rank sum test — Hochberg adjustment may be used; Median Difference (Net) = 0.24, 95% CI 2-sided [-0.01 to 0.96]
Statistical Analysis 5: Comparison: Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg vs Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg; Interleukin 6 (IL-6) at 3 weeks as compared to their respective baseline values; Test type: Other — Other: median difference; p = 0.055, Paired samples Wilcoxon rank sum test — Hochberg adjustment may be used; Median Difference (Net) = 0.39, 95% CI 2-sided [-0.03 to 4.61]
Statistical Analysis 6: Comparison: Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg vs Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg; Interleukin 6 (IL-6) at 5 weeks as compared to their respective baseline values; Test type: Other — Other: median difference; p = 0.06, Paired samples Wilcoxon rank sum test; Hochberg adjustment may be used; Median Difference (Net) = 0.54, 95% CI 2-sided [-0.06 to 1.96]
Statistical Analysis 7: Comparison: Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg vs Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg; Interleukin 8 (IL-8) at 3 weeks as compared to their respective baseline values; Test type: Other — Other: median difference; p = 0.420, Paired samples Wilcoxon rank sum test — Hochberg adjustment may be used; Median Difference (Net) = 0.73, 95% CI 2-sided [-1.63 to 1.62]
Statistical Analysis 8: Comparison: Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg vs Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg; Interleukin 8 (IL-8) at 5 weeks as compared to their respective baseline values; Test type: Other — Other: median difference; p = 0.733, Paired samples Wilcoxon rank sum test — Hochberg adjustment may be used; Median Difference (Net) = -0.39, 95% CI 2-sided [-1.315 to 1.31]
Statistical Analysis 9: Comparison: Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg vs Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg; Interleukin 10 (IL-10) at 3 weeks as compared to their respective baseline values; Test type: Other — Other: median difference; p = 0.010, Paired samples Wilcoxon rank sum test — Hochberg adjustment may be used; Median Difference (Net) = 0.12, 95% CI 2-sided [0.04 to 0.21]
Statistical Analysis 10: Comparison: Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg vs Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg; Interleukin 10 (IL-10) at 5 weeks as compared to their respective baseline values; Test type: Other — Other: median difference; p = 0.014, Paired samples Wilcoxon rank sum test — Hochberg adjustment may be used; Median Difference (Net) = 0.10, 95% CI 2-sided [0.04 to 0.40]

10. Secondary Outcome: Changes in the Immune Parameters Obtained From Biopsies
Description: All evaluable participants will have determinations of many immune parameters at baseline, 3 months, and 6 months. The changes in the parameters obtained from biopsies will be obtained from baseline vs. a single second biopsy at 6 months. Comparisons of the paired values will be performed using a Wilcoxon signed rank test, and a Hochberg adjustment may be used.
Time Frame: baseline, 3 months, and 6 months
Reporting Status: Not Posted, anticipated posting 2026-02

11. Secondary Outcome: Disease Free Survival (DFS)
Description: A DFS curve will be created using the Kaplan-Meier method based on all participants considered to be evaluable based on having received protocol treatment. DFS survival is defined as the time from the start of treatment until disease recurrence or death. Recurrence is suspected and/or determined by urine cytology and/or cystoscopic exam and then confirmed pathologically after a bladder biopsy or transurethral resection of bladder tumor (TURBT).
Time Frame: Assessed from start of therapy to disease recurrence or last follow up; up to 1 year.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Total Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg
Number analyzed (Participants) | 12 | 3 | 15
Weeks | 12.8 [12.3 to NA] — The upper Confidence Interval limit was NOT ACHIEVED/NEVER ATTAINED, i.e., CANNOT be calculated. There were not enough events for it to be determined. | 50.1 [12.3 to NA] — The upper Confidence Interval limit was NOT ACHIEVED/NEVER ATTAINED, i.e., CANNOT be calculated. There were not enough events for it to be determined. | 13.2 [12.28 to NA] — The upper Confidence Interval limit was NOT ACHIEVED/NEVER ATTAINED, i.e., CANNOT be calculated. There were not enough events for it to be determined.
Statistical Analysis 1: Comparison: Total Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg; Disease free survival time was evaluated with the product-limit estimator by Kaplan-Meier test; Test type: Other — One curve estimated in this cohort. Not compared to any other curves; Kaplan-Meier product-limit estimates — Unadjusted p-value; Kaplan-Meier product-limit = 13.2, 97.5% CI 2-sided [2.5 to 97.5]

12. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Through study completion, an average of 315 days.
Measure: Count of Participants; unit: Participants
Groups:
- Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg: Durvalumab 1500 mg is administered intravenously (IV) once every 4 weeks for 12 months with an option to continue therapy for an additional 12 months (total of 24 months) provided that patient is tolerating therapy and remains free of recurrent high grade non-muscle invasive bladder cancer (NMIBC) (see Treatment Period below). The dose of durvalumab is 1500 mg. If optional maintenance therapy continued in the second year, durvalumab 1500 mg will be administered intravenously once every 3 months to provide an immune boost.
  Vicineum is administered in a 12-week Induction Phase followed by a Maintenance Phase for at least one year with an option for a total of up to 2 years of treatment. During the Induction Phase, Vicineum is administered once weekly for 12 weeks. During the Maintenance Phase, Vicineum is administered every other week. The dose of Vicineum is 30 mg in 50 mL of saline.
- Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg: Durvalumab + Vicineum, at the maximum tolerated dose (MTD). Durvalumab: an option to continue therapy for an additional 12 months (total of 24 months) provided that participant is tolerating therapy and remains free of recurrent high grade NMIBC (see Treatment Period below). The dose of durvalumab is 1500 mg. If optional maintenance therapy continued in the second year, durvalumab 1500 mg will be administered intravenously once every 3 months to provide an immune boost.
  Vicineum is administered in a 12-week Induction Phase followed by a Maintenance Phase for at least one year with an option for a total of up to 2 years of treatment. During the Induction Phase, Vicineum is administered once weekly for 12 weeks. During the Maintenance Phase, Vicineum is administered every other week. The dose of Vicineum is 30 mg in 50 mL of saline.
Arm/Group | Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg
Number analyzed (Participants) | 12 | 3
Participants | 12 | 3

13. Other Pre Specified Outcome: Maximum Tolerated Dose (MTD) of Durvalumab
Description: The MTD will be identified based on being the dose level at which 0 or 1 participants in 6 has a dose-limiting toxicity (DLT). A DLT will be defined as any Grade 3 or higher toxicity that occurs during the initial 6-week period the subject is on treatment (i.e., the DLT evaluation period). Grade 3 is severe, grade 4 is life-threatening and grade 5 is death related to adverse event.
Time Frame: 6 weeks
Measure: Number; unit: Mg
Groups:
- All Participants: All participants that received durvalumab + vicineum in the run-in and expansion cohort.
Arm/Group | All Participants
Number analyzed (Participants) | 15
Mg | 1500

14. Other Pre Specified Outcome: Maximum Tolerated Dose (MTD) of Vicineum
Description: as for outcome 13
Time Frame: 6 weeks
Measure: Number; unit: Mg
Arm/Group | All Participants
Number analyzed (Participants) | 15
Mg | 30

15. Other Pre Specified Outcome: Dose-Limiting Toxicity (DLT)
Description: A DLT will be defined as any Grade 3 or higher toxicity that occurs during the initial 6-week period the subject is on treatment (i.e., the DLT evaluation period). Grade 3 is severe, grade 4 is life-threatening and grade 5 is death related to adverse event.
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg
Number analyzed (Participants) | 12 | 3
percentage of participants
  Grade 3 | 33.3 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 315 days
Arm/Group | Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg | Total Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/3 | 0/15
Serious Adverse Events (participants affected / at risk) | 4/12 | 0/3 | 4/15
Other Adverse Events (participants affected / at risk) | 12/12 | 3/3 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg (N=12) | Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg (N=3) | Total Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg (N=15)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-In Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg (N=12) | Expansion Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg (N=3) | Total Cohort - Durvalumab 1500mg Intravenous (IV) Every 4 Weeks (Q4WK) + Vicineum 30 mg (N=15)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 0 (0) | 2 (3)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 2 (2) | 0 (0) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Cardiac disorders - Other, Irregular heart rate (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 2 (2) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3)
Creatinine increased (Investigations) | 2 (2) | 2 (2) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 3 (3)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Eye disorders - Other, Hordeolum (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Eye disorders - Other, Ring of black string (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 2 (2) | 4 (4)
Fever (General disorders) | 1 (1) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Hematuria (Renal and urinary disorders) | 8 (8) | 0 (0) | 8 (8)
Hemoglobinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 3 (3)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 2 (2) | 0 (0) | 2 (2)
Malaise (General disorders) | 1 (1) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Left side pubic pressure (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Myalgia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 3 (10) | 1 (1) | 4 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0) | 5 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 3 (3)
Renal and urinary disorders - Other, Bilirubinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, Cloudy urine (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, Nitrite positive urine (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, UTI (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, decreased force of stream (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other, Penile itching (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 2 (2) | 0 (0) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, diffuse patchy rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, diffuse patchy skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 5 (5) | 0 (0) | 5 (5)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (3) | 0 (0) | 1 (3)
Urinary tract infection (Infections and infestations) | 5 (5) | 0 (0) | 5 (5)
Urinary urgency (Renal and urinary disorders) | 2 (4) | 0 (0) | 2 (4)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 2 (2) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-22): https://cdn.clinicaltrials.gov/large-docs/93/NCT03258593/Prot_SAP_002.pdf
  • Informed Consent Form (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT03258593/ICF_001.pdf